CLINICAL TRIAL: NCT01207050
Title: Pilot Study: The Effect of Rozerem on Sleep Disturbance After Traumatic Brain Injury
Brief Title: Effect of Rozerem on Sleep Among People With Traumatic Brain Injury
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Anthony Lequerica, Neuropsychologist and Clinical Research Scientist, Kessler Foundation
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: D-604-08; 10-3222-BIR-E-0 (Other Grant/Funding Number: New Jersey Commission on Brain Injury Research)
Record Dates: First submitted 2010-09-21; First posted 2010-09-22 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Insomnia; Brain Injury
Keywords: sleep disorders; traumatic brain injury
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Brain Injuries; Sleep Wake Disorders; Brain Injuries, Traumatic | interventions — ramelteon; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rozerem (Ramelteon) (Experimental): The primary drug of interest is a melatonin agonist for the treatment of insomnia.
  Interventions: Drug: Ramelteon
- Sugar pill (Placebo Comparator): Control condition.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Drug: Ramelteon — 8mg capsule taken within one half hour of bedtime each night over the three night study period.
  Other Names: Rozerem
  Arms: Rozerem (Ramelteon)
Dietary Supplement: Placebo — Control treatment
  Other Names: sugar pill
  Arms: Sugar pill

SUMMARY:
This pilot study proposes to examine the effect of Rozerem on sleep/wake patterns among individuals with Traumatic Brain Injury (TBI) experiencing sleep disturbance, using both objective and subjective measures. It will also show that improvement in sleep/wake patterns resulting from Rozerem will impact daytime functioning using objective and subjective measures.

DETAILED DESCRIPTION:
Although research has begun to examine sleep quality within the traumatic brain injury (TBI) population, most of the studies found in the research literature utilize subjective, self-report measures that can be problematic in terms of response accuracy when used with populations that have known cognitive deficits (Baños, LaGory, Sawrie, Faught, Knowlton, Prasad, Kuzniecky and Martin, 2004). Because TBI often results in a diminished capacity for self-reflective awareness, obtaining reliable sleep-related information is difficult to do through surveys alone (Fleming, Strong, Ashton, 1996; Vanderploeg, Belanger, Duchnick, and Curtiss, 2007).

A number of studies have attempted to objectify the measurement of sleep quality in TBI rehabilitation by having nursing staff keep an overnight log to document whether the patient was asleep or awake at hourly intervals (Burke, Shah, Schneider, Ahangar, & Al Aladai, 2004; Worthington & Melia, 2006). Because this results in only one single observation point per hour, it misses the nuances of the sleep/wake cycle obtained through more continuous measurement throughout the night and is still somewhat subjective and dependent on the observer's judgment.

Polysomnography, the electrophysiological measurement of sleep, is widely used in the clinical setting to diagnose sleep disorders. Using this more objective measure, Masel and colleagues (2001) found a high prevalence of posttraumatic hypersomnia, sleep apnea-hypopnea syndrome and periodic limb movement disorder that was not identified through self-report measures (Masel, Scheibel, Kimbark, & Kuna, 2001). This illustrates the limitations of self-report questionnaires and highlights the need for more objective measures. However, the high cost and inconvenience of polysomnography, requiring multiple electrodes attached to the face, head, and other parts of the body, make it less practical for research studies.

These limitations of subjective self-report measures and the cost and inconvenience of polysomnography suggest the need for alternative methods of measurement. With the use of an actigraph, a small, highly sensitive, accelerometer (motion detector) worn on the wrist over a period of days, a number of sleep-related variables can be derived through the analysis of motion and rest patterns using a computer algorithm (Coffield & Tryon, 2004). Variables such as sleep latency, total time asleep, and number of nocturnal awakenings derived through actigraphy are comparable to those obtained via polysomnography, and recent research studies demonstrate the validity of actigraph-based sleep/wake estimates among individuals with acquired brain injury (Muller, Czymmek, Thone-Otto, & Von Cramon, 2006; Tweedy & Trost, 2005; Schuiling, Rinkel, Walchenbach, & de Weerd, 2005). Thus, actigraphy represents a means of measurement that will enable the collection of objective data in the comfort of the sleeper's usual environment in a manner that is less invasive and more cost-effective than polysomnography, and more reliable than self-report measures alone.

The most widely researched treatments for sleep disturbance are problematic for individuals with TBI due to their effects on cognition and risk for dependence. With a high prevalence of sleep/wake disorders found among individuals with TBI, Rozerem is a promising treatment option to improve sleep quality that is less likely to exacerbate cognitive sequelae of TBI and less likely to result in dependence.

ELIGIBILITY:
Inclusion Criteria:

1. History of traumatic brain injury (TBI) as determined by any of the following at least 1 month prior to study entry:

   * Glasgow Coma Scale Score < 15
   * Loss of consciousness greater than 5 minutes
   * Post traumatic amnesia greater than 30 minutes
   * Abnormal neuro-imaging findings after TBI
   * Evidence of neurologic deficit as a result of TBI
2. Endorsement of any of the following by self-report or proxy-report:

   * Problems falling or staying asleep
   * Daytime sleepiness or fatigue (either cognitive or physical)
   * These symptoms must be identified as having an onset after TBI
   * Score of > 5 on the Pittsburgh Sleep Quality Index (PSQI)
3. Typical bedtime between 8pm and midnight with wake-up time between 6am and 10am on weekdays.
4. Must be living in the community
5. In the opinion of the Study Team, the participant must be deemed reliable and likely to make all study visits

Exclusion Criteria:

1. Bilateral arm fractures, cellulitis or other conditions that prevent safe wearing of the actigraph
2. Individuals using other known hypnotic agents (i.e., benzodiazepines, diphenhydramine, zolpidem) will be considered for participation but must have refrained from using sleep medication for two weeks prior to the study and throughout the course of the study
3. Movement disorder or spasticity affecting both upper extremities
4. Severe pain or history of chronic pain
5. Individuals with multiple musculoskeletal injuries
6. Taking luvox or fluvoxamine (medication that potentially interact with ramelteon
7. Liver disease
8. Patients who are ventilator-dependent
9. Penetrating head TBI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-09; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Sleep Quality | At third week of treatment
  Sleep Latency (the number of minutes it takes for the participant to fall asleep after getting into bed), and Total Sleep Time (number of minutes asleep between getting into bed for the night and getting out of bed in the morning).

SECONDARY OUTCOMES:
Epworth Sleepiness Scale | After completing two weeks of treatment
  Measure of subjective daytime sleepiness.
Cognitive Performance | After completing two weeks of treatment
  Performance on a computer-administered continuous performance test.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Lequerica, PhD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation Research Center, West Orange, New Jersey, United States

REFERENCES:
- [Background] Banos JH, LaGory J, Sawrie S, Faught E, Knowlton R, Prasad A, Kuzniecky R, Martin RC. Self-report of cognitive abilities in temporal lobe epilepsy: cognitive, psychosocial, and emotional factors. Epilepsy Behav. 2004 Aug;5(4):575-9. doi: 10.1016/j.yebeh.2004.04.010. PMID 15256196
- [Background] Fleming JM, Strong J, Ashton R. Self-awareness of deficits in adults with traumatic brain injury: how best to measure? Brain Inj. 1996 Jan;10(1):1-15. doi: 10.1080/026990596124674. PMID 8680388
- [Background] Vanderploeg RD, Belanger HG, Duchnick JD, Curtiss G. Awareness problems following moderate to severe traumatic brain injury: Prevalence, assessment methods, and injury correlates. J Rehabil Res Dev. 2007;44(7):937-50. doi: 10.1682/jrrd.2006.12.0163. PMID 18075951
- [Background] Burke DT, Shah MK, Schneider JC, Ahangar B, Al Aladai S. Sleep-wake patterns in brain injury patients in an acute inpatient rehabilitation hospital setting. The Journal of Applied Research 4(2):239-244, 2004.
- [Background] Worthington AD, Melia Y. Rehabilitation is compromised by arousal and sleep disorders: results of a survey of rehabilitation centres. Brain Inj. 2006 Mar;20(3):327-32. doi: 10.1080/02699050500488249. PMID 16537274
- [Background] Masel BE, Scheibel RS, Kimbark T, Kuna ST. Excessive daytime sleepiness in adults with brain injuries. Arch Phys Med Rehabil. 2001 Nov;82(11):1526-32. doi: 10.1053/apmr.2001.26093. PMID 11689971
- [Background] Coffield TG, Tryon WW. Construct validation of actigraphic sleep measures in hospitalized depressed patients. Behav Sleep Med. 2004;2(1):24-40. doi: 10.1207/s15402010bsm0201_3. PMID 15600222
- [Background] Muller U, Czymmek J, Thone-Otto A, Von Cramon DY. Reduced daytime activity in patients with acquired brain damage and apathy: a study with ambulatory actigraphy. Brain Inj. 2006 Feb;20(2):157-60. doi: 10.1080/02699050500443467. PMID 16421064
- [Background] Schuiling WJ, Rinkel GJ, Walchenbach R, de Weerd AW. Disorders of sleep and wake in patients after subarachnoid hemorrhage. Stroke. 2005 Mar;36(3):578-82. doi: 10.1161/01.STR.0000154862.33213.73. Epub 2005 Jan 27. PMID 15677579
- [Background] Tweedy SM, Trost SG. Validity of accelerometry for measurement of activity in people with brain injury. Med Sci Sports Exerc. 2005 Sep;37(9):1474-80. doi: 10.1249/01.mss.0000177584.43330.ae. PMID 16177597
- See also: Click here for further information about this study — http://www.kesslerfoundation.org